CLINICAL TRIAL: NCT03183895
Title: Safety and Performance Evaluation of the AccuCinch® Ventricular Restoration System for the Treatment of Heart Failure With or Without Functional Mitral Regurgitation Due to Dilated Ischemic or Non-Ischemic Cardiomyopathy - The CorCinch-EU Study
Brief Title: Evaluate the Safety and Performance of the AccuCinch® Ventricular Repair System - The CorCinch-EU Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4631
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure; Cardiomyopathies
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Left ventricular restoration — The AccuCinch® Ventricular Repair System, implanted in the sub-valvular space of the left ventricle, is intended to reduce significant symptomatic mitral regurgitation and reverse left ventricular remodeling due to dilated cardiomyopathy of either ischemic or non-ischemic etiology via percutaneous interventional methods.

SUMMARY:
This is prospective, non-randomized, single-arm, international, multicenter, clinical safety and performance clinical investigation to evaluate the AccuCinch® Ventricular Repair System for the treatment of heart failure, with or without functional mitral regurgitation due to dilated ischemic or non-ischemic cardiomyopathy

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate the safety and performance of the AccuCinch Ventricular Repair System for the treatment of heart failure and functional mitral regurgitation in symptomatic adult patients with or without functional mitral regurgitation (FMR) and left ventricular remodeling due to dilated cardiomyopathy (ischemic or non-ischemic etiology), who remain symptomatic despite optimized medical therapy.

Subjects with FMR must present with at least moderate FMR, a reduced ejection fraction (≤40%) and high operative risk as assessed by the Heart Team. The Heart Team may utilize established risk scores (STS, Euro-Score II) in conjunction with comorbidities as recommended by MVARC (frailty index; major organ system compromise not to be improved postoperatively; procedure specific impediments).

Subjects without FMR must present a markedly dilated left ventricle with LVEDD ≥ 55 mm and reduced ejection fraction (≤40%). These patients are not potential candidates for "conventional intervention", because their mitral valve is not in need of repair or replacement. Therefore, AccuCinch represents the sole treatment option for these patients, who are not selected on the basis of high surgical risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Subjects who present with heart failure with or without functional mitral regurgitation due to dilated cardiomyopathy of ischemic or non-ischemic etiology

  1. For subjects with FMR, severity of FMR: ≥ Moderate 2+
  2. For subjects without FMR, LVEDD ≥ 55 mm
* Ejection Fraction: ≥20 to ≤40%
* Symptom Status: NYHA II-IVa
* Patients to be considered for the present study will be required to have received all appropriate guidelines-recommended therapies for at least 3 months prior to the enrollment with stable doses of drugs for at least 1 month.
* Surgical risk:

  1. For patients with FMR only: the Heart Team must assess as high-risk and may utilize risk score or comorbidities to demonstrate high risk features. High risk for mitral valve surgery is defined utilizing established risk scores (STS, Euro-Score II) in conjunction with comorbidities as recommended by MVARC (frailty index; major organ system compromise not to be improved postoperatively; procedure specific impediments) (MVARC Part 1)
  2. For all patients: Subject is eligible for cardiac surgery (namely, the patient is in a condition that allows a potential conversion to open surgery in case of procedural complications). This criterion adds a safety level for the patients
* Completion of all qualifying diagnostic and functional tests and agrees to comply with study follow-up schedule
* Patients required to have an ICD are required to have ICD implant at least 1 month prior to enrollment

Exclusion Criteria:

* Life expectancy <1 yr due to noncardiac conditions
* NYHA functional class IVb or ACC/AHA stage D heart failure
* Hypotension (systolic pressure <90 mm Hg) or requirement for inotropic support or mechanical hemodynamic support
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or nonischemic etiology
* Fixed pulmonary artery systolic pressure >70 mm Hg
* Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction
* Mitral valve anatomy which may preclude proper device treatment
* Mitral valve area <4.0 cm2 (if new device therapy may further decrease the mitral orifice area)
* Any prior mitral valve surgery or transcatheter mitral valve procedure
* Stroke or transient ischemic event within 30 days
* Modified Rankin Scale ≥ 4 disability
* Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months
* Untreated clinically significant coronary artery disease requiring revascularization
* Severe symptomatic carotid stenosis (>70% by ultrasound).
* Myocardial infarction ≤ 30 days
* Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days
* Tricuspid valve disease requiring surgery or severe tricuspid regurgitation (per ASE guidelines; core lab assessment)
* Aortic valve disease requiring surgery
* Moderate or severe aortic valve stenosis or regurgitation
* Aortic valve prosthesis
* Fluoroscopic or echocardiographic evidence of severe aortic arch calcification, mobile aortic atheroma, intracardiac mass, thrombus, or vegetation
* Need for any cardiovascular surgery (other than for MV disease)
* Active endocarditis
* Anatomical pathology/constraints preventing appropriate access/implant of the AccuCinch System (e.g., femoral arteries will not support an 20F system)
* Known allergy to nickel, polyester, or polyethylene
* Active infections requiring current antibiotic therapy
* Subjects in whom transesophageal echocardiography is contraindicated
* Renal insufficiency (i.e., eGFR of <30ml/min/1.73m2; Stage 4 or 5 CKD)
* Subjects in whom anticoagulation or antiplatelet therapy is contraindicated
* Any prior true anaphylactic reaction to contrast agents; defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to procedure.
* Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter defibrillator within 1 month
* Absence of CRT with class I indication criteria for biventricular pacing (left bundle branch block pattern and QRS duration ≥150 ms)
* Subjects on high dose steroids or immunosuppressant therapy
* Any condition making it unlikely the patient will be able to complete all protocol procedures (including compliance with guideline directed medical therapy) and follow-up visits
* Patient is unable or unwilling to sign written patient information sheet and informed consent form before study enrollment. This study excludes vulnerable populations as defined in protocol section 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety outcome: 30-day major adverse events (MAEs) | 30-day
  Major adverse event (MAE) where MAE is a composite of the following device- or procedure-related events:
  A. All-cause mortality
  B. Stroke
  C. Life-threatening bleeding (MVARC scale)
  D. Major vascular complications
  E. Major cardiac structural complications
  F. Myocardial infarction or coronary ischemia requiring PCI or CABG
  G. Stage 2 or 3 acute kidney injury (includes new dialysis)
  H. Severe hypotension, worsening of heart failure, or respiratory failure requiring intravenous pressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for >48 h.
  I. Emergency surgery or re-intervention related to the device or access procedure

SECONDARY OUTCOMES:
Technical success: Successful access, delivery, and retrieval of AccuCinch System components, successful deployment of the AccuCinch implant without need for unplanned or emergency surgery or re-intervention | 30-day
  Successful access, delivery, and retrieval of all AccuCinch catheters. Deployment and correct positioning of the intended AccuCinch implant, and no need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure measured upon completion of the procedure.
Structural performance: Assessment of device integrity | 30-day
  No migration, embolization, detachment, fracture, hemolysis, thrombosis or endocarditis; and no para-device complications (erosion, effusion requiring surgery or drainage or producing tamponade, damage to the MV apparatus)
Clinical outcome: Freedom from re-hospitalizations or re-interventions for the underlying condition | 30-day
  Freedom from re-hospitalizations or re-interventions for the underlying condition
Clinical outcome: Improvement in NYHA functional class | 30-day
  Improvement in NYHA functional class when compared to baseline assessment
Clinical outcome: Improvement in six-minute walk test | 30-day
  Improvement in six-minute walk test (6MWT) when compared to baseline assessment
Clinical outcome: Improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) Quality of Life (QoL) | 30-day
  Improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) Quality of Life (QoL) when compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, CCRA, Study Director — Ancora Heart, Inc.
Locations (19):
- Republican Scientific and Practical Centre of Cardiology, Minsk, Belarus
- Belgium (2):
  - Onze Lieve Vrouwziekenhuis, Aalst, Aaslt
  - AZ Sint-Jan Brugge, Bruges
- Na Homolce Hospital, Prague, Czechia
- France (6):
  - Pessac (CHU Bordeaux), Pessac, Avenue Magellen
  - Hôpital Cardio-Vasculaire Louis Pradel, Bron
  - Hôpital de La Timone, Marseille
  - Paris Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Civil de Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse
- Italy (3):
  - IRCCS Policlinico San Donato, Milan, Piazza Edmondo Malan, 1 San Donato Milanese,
  - Maria Cecilia Hospital, Cotignola, Via Madonna Di Genova, 1,
  - Ospedale San Raffaele, Milan, Via Olgettina, 60,
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
- Medical University of Warsaw, Warsaw, Poland
- University Hospital Zurich, Zurich, Switzerland
- Royal Brompton & Harefield NHS Trust, London, Sydney St, Chelsea, London, United Kingdom